CLINICAL TRIAL: NCT02807103
Title: Evaluation of Rituximab-based Regimen Compared to Conventional Therapeutic Strategy For Remission Induction In Patients With Newly-Diagnosed or Relapsing Eosinophilic Granulomatosis With Polyangiitis. Prospective, Randomized, Controlled, Double-blind Study
Brief Title: Rituximab in Eosinophilic Granulomatosis With Polyangiitis
Acronym: REOVAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Vasculitis Study Group (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P140915; 2016-000275-25 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-06-21 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis (EGPA)
Keywords: Rituximab; remission induction; eosinophilic granulomatosis with polyangiitis
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — Rituximab; Sodium Chloride; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rituximab with FFS=0 (Experimental): All patients in the rituximab group will receive corticosteroids with a predefined tapering schedule similar to the conventional therapy group.
  Patients with FFS=0 will receive 1 gram of rituximab at day 1 and day 15 as induction treatment
  Interventions: Drug: Rituximab
- Conventional therapy with FFS=0 (Placebo Comparator): All patients will receive corticosteroids with a predefined tapering schedule similar to the experimental group.
  Patients with FFS=0 will receive placebo-rituximab at day 1 and day 15.
  Interventions: Drug: Placebo-rituximab
- Rituximab with FFS≥1 (Experimental): All patients in the rituximab group will receive corticosteroids with a predefined tapering schedule similar to the conventional therapy group.
  Patients with FFS≥1 will receive a total of 9 pulses :
  * 1 gram of rituximab at day 1 and day 15 as induction treatment
  * placebo-cyclophosphamide at days 1, 15, 29, 50, 71, 92, 113, 134 and 155.
  Maintenance therapy by azathioprine will be started at day 180 according to the standard of care of these patients, as recommended by the French Vasculitis Study Group.
  Interventions: Drug: Rituximab; Drug: Placebo-cyclophosphamide
- Conventional therapy with FFS≥1 (Active Comparator): All patients will receive corticosteroids with a predefined tapering schedule similar to the experimental group.
  Patients with FFS≥1 will receive intravenous pulses of cyclophosphamide for a total of 9 pulses: 600 mg/m2 at days 1, 15 and 29, and then 500 mg-fixed dose at days 50, 71, 92, 113, 134 and 155.
  Maintenance therapy by azathioprine will be started at day 180 according to the standard of care of these patients, as recommended by the French Vasculitis Study Group.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rituximab — 1 g intravenous pulse at day1 and day15
  Other Names: Mabthera
  Arms: Rituximab with FFS=0; Rituximab with FFS≥1
Drug: Placebo-rituximab — intravenous pulses at day1 and day15
  Other Names: nacl
  Arms: Conventional therapy with FFS=0
Drug: Cyclophosphamide — intravenous 9 pulses : 600 mg/m2 at days 1, 15 and 29, and then 500 mg-fixed dose at days 50, 71, 92, 113, 134 and 155.
  Other Names: endoxan
  Arms: Conventional therapy with FFS≥1
Drug: Placebo-cyclophosphamide — intravenous 7 pulses : at days 29, 50, 71, 92, 113, 134 and 155.
  Other Names: Nacl
  Arms: Rituximab with FFS≥1

SUMMARY:
Phase III, comparative, multicenter, randomized, controlled, double-blind and superiority research, comparing rituximab-based regimen with conventional therapeutic strategy for the induction of remission in patients with eosinophilic granulomatosis with polyangiitis (EGPA).

Patients with newly diagnosed or relapsing EGPA will be randomized in a 1:1 ratio to receive:

* Experimental therapeutic strategy based on the use of rituximab (experimental group)
* Conventional therapeutic strategy based on Five-Factor Score (FFS)-assessed disease severity (comparative group)

DETAILED DESCRIPTION:
Systemic vasculitides are inflammatory diseases of blood vessels, among which anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV) are often severe with life-threatening manifestations or complications. AAV include granulomatosis with polyangiitis (GPA), microscopic polyangiitis (MPA) and eosinophilic granulomatosis with polyangiitis (EGPA, formerly Churg-Strauss syndrome).

Cytotoxic drugs and glucocorticoids have been the standard of care for remission induction for nearly five decades. This regimen improved the outcome of severe AAV from death to a strong likelihood of disease control and temporary remission. However, a remission is not obtained in all patients with this combination of drugs, and most patients experience disease flares requiring repeated treatment with associated significant morbidity and mortality.

In 2 prospective controlled trials, rituximab, an anti-CD20 monoclonal antibody, was shown to be non inferior to cyclophosphamide to induce remission with an acceptable safety profile in patients with systemic GPA and MPA. However, patients with EGPA were not included in these trials and rituximab has not been evaluated prospectively to induce remission in this disease which pathogenesis is complex and not only restricted to ANCA responsibility.

In patients with EGPA, overall survival is good when treatment is stratified according to prognostic factors (Five Factor Score) but long-term outcome is not so good since relapses occur in more than 40% of patients, leading to high cumulative morbidity and damage. In small retrospective studies, rituximab seems promising as a remission-induction agent in patients with EGPA, independently from the ANCA status.

The trial detailed here is the first prospective trial evaluating rituximab as induction-remission treatment for EGPA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of EGPA independently of ANCA status,
* Patient aged of 18 years or older,
* Patients with newly-diagnosed disease or relapsing disease at the time of screening, with an active disease defined as a Birmingham Vasculitis Activity Score (BVAS) ≥3,
* Patients within the first 21 days following initiation/increase of corticosteroids at a dose ≤ 1 mg/kg/day (pulses of methylprednisolone before oral corticosteroid therapy are authorized) ,
* Patient able to give written informed consent prior to participation in the study.

Exclusion Criteria:

* Patients with GPA, MPA, or other vasculitides, defined by the ACR criteria and/or the Chapel Hill Consensus Conference,
* Patients with vasculitis in remission of the disease defined as a BVAS <3,
* Patients with severe cardiac failure defined as class IV in New York Heart Assocation
* Patients with acute infections or chronic active infections (including HIV, HBV or HCV),
* Patients with active cancer or recent cancer (<5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment,
* Pregnant women and lactation. Patients with childbearing potential should have reliable contraception for the 12 months duration of the study,
* Patients with EGPA who have already been treated with rituximab within the previous 12 months,
* Patients with hypersensitivity to a monoclonal antibody or biologic agent,
* Patients with contraindication to use rituximab, cyclophosphamide, mesna or azathioprine,
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patients included in other investigational therapeutic study within the previous 3 months,
* Patients suspected not to be observant to the proposed treatments,
* Patients who have white blood cell count ≤4,000/mm3,
* Patients who have platelet count ≤100,000/mm3,
* Patients who have ALT or AST level greater that 3 times the upper limit of normal that cannot be attributed to underlying EGPA disease,
* Patients unable to give written informed consent prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who obtained a BVAS=0 and prednisone dose ≤7.5 mg/day at day 180. | 180 days

SECONDARY OUTCOMES:
Number of adverse events | 180 days
  expressed as adverse events according to the CTCAE toxicity grading system per patient-year for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, hemorrhagic cystitis, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions
Number of adverse events | 360 days
  expressed as adverse events according to the CTCAE toxicity grading system per patient-year for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, hemorrhagic cystitis, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions
Area under the curve for corticosteroids | 180 days
  To measure the corticosteroid dose and to compare the corticosteroid sparing effect of rituximab versus conventional therapy
Area under the curve for corticosteroids | 360 days
  To measure the corticosteroid dose and to compare the corticosteroid sparing effect of rituximab versus conventional therapy
Number of sequelae assessed by the Vasculitis Damage Index | 180 days
Number of sequelae assessed by the Vasculitis Damage Index | day 180 and day 360
ANCA titers and CD19+cells | day 180 and day 360
Health Assessment Questionnaire (HAQ) score | 180 days
  to evaluate functional disability
Health Assessment Questionnaire (HAQ) score | 360 days
  to evaluate functional disability
Short Form-36 score | 180 days
  to evaluate quality of life
Short Form-36 score | 360 days
  to evaluate quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PUECHAL, MD, PhD, Study Chair — Centre de référence " Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques "
Locations (1):
- Hôpital Cochin, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Terrier B, Pugnet G, de Moreuil C, Bonnotte B, Benhamou Y, Chauveau D, Besse MC, Duffau P, Limal N, Neel A, Urbanski G, Jourde-Chiche N, Martin-Silva N, Campagne J, Mekinian A, Schleinitz N, Ackermann F, Fauchais AL, Froissart A, Le Gallou T, Uzunhan Y, Viallard JF, Berezne A, Chiche L, Taille C, Direz G, Durel CA, Godmer P, Trad S, Lambert M, de Menthon M, Quemeneur T, Cadranel J, Charles P, Dossier A, Jilet L, Guillevin L, Abdoul H, Puechal X; French Vasculitis Study Group. Rituximab Versus Conventional Therapy for Remission Induction in Eosinophilic Granulomatosis With Polyangiitis : A Randomized Controlled Trial. Ann Intern Med. 2025 Sep;178(9):1249-1257. doi: 10.7326/ANNALS-24-03947. Epub 2025 Jul 29. PMID 40720835
- See also: Related Info — http://www.vascularites.org/